CLINICAL TRIAL: NCT05216991
Title: The Role of Sugammadex and Quantitative Monitoring in "Fast-Track Anesthesia" During Liver Transplantation
Brief Title: Sugammadex and Quantitative Monitoring in "Fast-Track Anesthesia" During Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, J. Ross Renew, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 21-011838
Record Dates: First submitted 2022-01-19; First posted 2022-02-01 (Actual); Results first posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-09

CONDITIONS: Liver Transplant Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TetraGraph monitoring on dominant hand: Patients receiving sugammadex after undergoing liver transplantation with quantitative monitoring as standard of care
  Interventions: Other: TetraGraph on dominant hand
- TetraGraph monitoring on non-dominant hand: Patients receiving sugammadex after undergoing liver transplantation with quantitative monitoring as standard of care
  Interventions: Other: TetraGraph on non-dominant hand

INTERVENTIONS:
Other: TetraGraph on dominant hand — Using standard of care TetraGraph device on dominant hand
  Groups: TetraGraph monitoring on dominant hand
Other: TetraGraph on non-dominant hand — Using standard of care TetraGraph device on non-dominant hand
  Groups: TetraGraph monitoring on non-dominant hand

SUMMARY:
The purpose of this research is to estimate the frequency of postoperative lasting muscle weakness in patients receiving Sugammadex after undergoing liver transplant surgery by using electromyographic device (EMG), such as TetraGraph.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to participate and provide an informed consent.
* Patients undergoing primary liver transplantation.

Exclusion Criteria:

* Patients with unilateral disorders, such as stroke, carpal tunnel syndrome, broken wrist with nerve damage, Dupuytren contracture, or any similar wrist injury.
* Patients with systemic neuromuscular diseases such as myasthenia gravis.
* Patients with a known history of cerebrovascular accident (CVA).
* Patients undergoing repeat liver transplantation or concomitant pancreas/kidney transplantation at the time of liver transplantation.
* Patients admitted to the intensive care unit prior to liver transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing liver transplant surgery at Mayo Clinic in Florida. All study participants will receive their routine standard of care intraoperatively which consists of receiving sugmmadex as part of anesthesia, as well as, monitored with a quantitative monitor device on their dominant or nondominant hand, per standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Ross Renew, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 67 participants screen failed prior to randomization.
Groups:
- TetraGraph monitoring on dominant hand: Patients who received sugammadex after undergoing liver transplantation with quantitative monitoring as standard of care
  TetraGraph on dominant hand: Using standard of care TetraGraph device on dominant hand
- TetraGraph monitoring on non-dominant hand: Patients who received sugammadex after undergoing liver transplantation with quantitative monitoring as standard of care
  TetraGraph on non-dominant hand: Using standard of care TetraGraph device on non-dominant hand
Period: Overall Study
Arm/Group | TetraGraph monitoring on dominant hand | TetraGraph monitoring on non-dominant hand
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TetraGraph monitoring on dominant hand | TetraGraph monitoring on non-dominant hand | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (8.2) | 57.9 (7.5) | 57.0 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 11 | 9 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 15 | 12 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 15 | 14 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Postoperative Residual Weakness in the Recovery Room
Description: Number of patients to experience postoperative residual weakness after receiving Sugammadex as standard of care for liver transplant surgery. Postoperative residual weakness is defined as train-of-four ratio (TOF) <0.9. Train-of-four is a test used to measure the level of neuromuscular blockage through delivery of four consecutive stimuli to a nerve. Measurement of the muscle's response (number of twitches 1-4) to the stimuli indicates the degree of paralysis. This is measured by an EMG device placed on the thumb which is also part of standard of care for intraoperative assessment of muscle weakness. The ratio is calculated by comparing the amplitude of the fourth twitch to the first twitch. A TOF <0.9 indicates residual weakness, a TOF equal to or greater than 0.9 indicates no residual weakness.
Time Frame: Approximately 10 minutes of surgery recovery period
Measure: Count of Participants; unit: Participants
Arm/Group | TetraGraph monitoring on dominant hand | TetraGraph monitoring on non-dominant hand
Number analyzed (Participants) | 15 | 15
Participants | 2 | 0

2. Secondary Outcome: ICU Admission
Description: Number of patients to require ICU admission following liver transplantation
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | TetraGraph monitoring on dominant hand | TetraGraph monitoring on non-dominant hand
Number analyzed (Participants) | 15 | 15
Participants | 2 | 0

3. Secondary Outcome: Hospital Length of Stay
Description: Average number of days patients are admitted to the hospital following liver transplantation
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | TetraGraph monitoring on dominant hand | TetraGraph monitoring on non-dominant hand
Number analyzed (Participants) | 15 | 15
days | 6.1 (3.2) | 6.4 (2.4)

4. Secondary Outcome: Postoperative Pulmonary Complications
Description: Number of participants who experienced postoperative pulmonary complications defined as pneumonia and respiratory failure
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | TetraGraph monitoring on dominant hand | TetraGraph monitoring on non-dominant hand
Number analyzed (Participants) | 15 | 15
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through study completion, approximately 30 days.
Description: Adverse events were collected through specific questioning and/or examination.
Arm/Group | TetraGraph monitoring on dominant hand | TetraGraph monitoring on non-dominant hand
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 2/15 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TetraGraph monitoring on dominant hand (N=15) | TetraGraph monitoring on non-dominant hand (N=15)
Postoperative Residual Weakness (Musculoskeletal and connective tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT05216991/Prot_SAP_000.pdf